CLINICAL TRIAL: NCT01812525
Title: Moderate to Severe Bronchiolitis: Standard Therapy Versus Therapy With NaCl 3%
Brief Title: Moderate to Severe Bronchiolitis: Standard Therapy Versus Therapy With NaCl 3% Inhalations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Raphaelle Jaquet-Pilloud (Other)
Collaborators: Swiss Foundation for the Health of Children and Adolescents (Other)
Responsible Party: Sponsor-Investigator, Raphaelle Jaquet-Pilloud, Jean-Yves Pauchard, MD, Hôpital de L'Enfance
Organization: Hôpital de L'Enfance (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 453/12
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Moderate to Severe Bronchiolitis
Keywords: Bronchiolitis; Moderate to Severe; Hypertonic saline; NaCl 3% inhalations; Standard therapy; Wang score; in-patients
MeSH Terms: conditions — Bronchiolitis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NaCl 3% inhalations + standard therapy (Active Comparator): In this group, patients receive NaCl 3% inhalations ( 4ml QID) together with standard therapy.
  Standard therapy includes suctioning nasal secretions, water-electrolyte balance maintenance and oxygen supplementation when needed.
  Interventions: Drug: NaCl 3%; Other: Standard therapy
- Standard therapy (Placebo Comparator): Standard therapy includes suctioning nasal secretions, water-electrolyte balance maintenance and oxygen supplementation when needed
  Interventions: Other: Standard therapy

INTERVENTIONS:
Drug: NaCl 3% — NaCl 3%: 4ml QID
  Other Names: Mucoclear 3%
  Arms: NaCl 3% inhalations + standard therapy
Other: Standard therapy — Standard therapy includes suctioning nasal secretions, water-electrolyte balance maintenance and oxygen supplementation when needed

SUMMARY:
Our study will investigate inhalation therapy of NaCl 3% compared to standard therapy with no inhalation in the treatment of moderate to severe bronchiolitis. The impact on length of hospital stay will be analyzed.

DETAILED DESCRIPTION:
Acute viral bronchiolitis is the most common lower respiratory tract infection in the first year of life and leads to a large number of hospital admissions. The only recommended treatment is supportive. However many different types of drug inhalations have been studied but their efficacy remains controversial.

Our study will compare recommended supportive therapy to supportive therapy combined to hypertonic saline (NaCl 3%) inhalations in the treatment of moderate to severe bronchiolitis. This will be the first study to use a true control group with no inhalation.

ELIGIBILITY:
Inclusion Criteria:

* children between ages 6 weeks to 24 months
* first episode of wheezing
* diagnosis of moderate to severe bronchiolitis: The patients are ranked as moderately to severely ill according to the Wang clinical severity score

Exclusion Criteria:

* Children with mild bronchiolitis (Wang score < 5)
* Children with pre-existent cardiac disease
* Children with clinically significant chronic respiratory disease
* Immunocompromised children
* Children with a gestational age at birth less than 34 weeks
* Children who received immunoprophylaxis therapy (i.e RSV immune globulin therapy)
* Children who received corticosteroid in any form in the preceding 2 weeks before presentation
* Children who received bronchodilators within 24 hours before presentation
* Children with critical illness at presentation requiring immediate admission to intensive care unit

Ages: 6 Weeks to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2013-03; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 2 years
  The length of stay is defined as the time between study entry and the time at which the child reach protocol-defined discharge criteria as measured by the physician in charge.

SECONDARY OUTCOMES:
transfer rate to ICU | 2 years
readmission rate in the next 7 days following discharge | 2 years
Wang clinical severity score evolution | 2 years
adverse events | 2 years
Patients' ability to feed | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Pauchard, Study Director — Hôpital de l'Enfance, Lausanne, Switzerland
Locations (1):
- Hôpital de l'Enfance, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Jaquet-Pilloud R, Verga ME, Russo M, Gehri M, Pauchard JY. Nebulised hypertonic saline in moderate-to-severe bronchiolitis: a randomised clinical trial. Arch Dis Child. 2020 Mar;105(3):236-240. doi: 10.1136/archdischild-2019-317160. Epub 2019 Sep 5. PMID 31488402